CLINICAL TRIAL: NCT01197534
Title: (OSKIRA-2): A Phase III, Multi-centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study of Two Dosing Regimens of Fostamatinib Disodium in Rheumatoid Arthritis Patients With an Inadequate Response to DMARDs
Brief Title: Evaluation of Effectiveness of Two Dosing Regimens of Fostamatinib Compared to Placebo in Patients With Rheumatoid Arthritis (RA) Who Are Taking Disease Modifying Anti-rheumatic Drug (DMARD) But Not Responding.
Acronym: OSKIRA - 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00002; 2010-020744-35 (EudraCT Number)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dosing Regimen A (Experimental): Oral Treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen B (Experimental): Oral Treatment
  Interventions: Drug: fostamatinib
- Dosing Regimen C (Placebo Comparator): Oral Treatment
  Interventions: Drug: placebo, fostamatinib

INTERVENTIONS:
Drug: fostamatinib — fostamatinib 100 mg twice daily
  Arms: Dosing Regimen A
Drug: fostamatinib — fostamatinib 100 mg twice daily/ 150 mg once daily
  Arms: Dosing Regimen B
Drug: placebo, fostamatinib — Placebo for 24 weeks followed by fostamatinib 100 mg twice daily.
  Arms: Dosing Regimen C

SUMMARY:
The purpose of the study is to evaluate the effectiveness of two dosing regimens of fostamatinib compared to placebo, in patients with rheumatoid arthritis (RA) who are taking disease modifying anti-rheumatic drug (DMARD) but not responding. The study will last for 1 year.

DETAILED DESCRIPTION:
Sub-study:

Full title: Optional Genetic Research

Date: 18 June 2010

Version: 1

Objectives: To collect and store, with appropriate consent ,DNA samples for future exploratory research into genes/genetic variation that may influence response (ie, absorption, distribution, metabolism and excretion, safety, tolerability and efficacy) to fostamatinib disodium and/or methotrexate; and/or susceptibility to, progression of and prognosis of RA

ELIGIBILITY:
Inclusion Criteria:

* Active rheumatoid arthritis (RA) diagnosed after the age of 16
* Treatment with one the following disease modifying anti-rheumatic drug: methotrexate, sulfasalazine, hydroxychloroquine or chloroquine
* 4 or more swollen joints and 4 or more tender/painful joints (from 28 joint count)and either Erythrocyte Sedimentation Rate (ESR) blood result of 28mm/h or more, or C-Reactive Protein (CRP) blood result of 10mg/L or more
* At least one of the following: documented history of positive rheumatoid factor (blood test), current presence of rheumatoid factor (blood test), radiographic erosion within 12 months prior to study enrolment, presence of serum anti-cyclic citrullinated peptide antibodies (blood test)

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Poorly controlled hypertension
* Liver disease or significant liver function test abnormalities
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders
* Recent or significant cardiovascular disease
* Significant active or recent infection including tuberculosis
* Previous failure to respond to a TNF alpha antagonist, anakinra or previous treatment with other biological agent
* Severe renal impairment
* Neutropenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil MacKillop, MD PhD, Study Director — AstraZeneca
Locations (149):
- United States (57):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Huntington Beach, California
  - Research Site, Torrance, California
  - Research Site, Trumbull, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Venice, Florida
  - Research Site, Zephyrhills, Florida
  - Research Site, Canton, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Boise, Idaho
  - Research Site, South Bend, Indiana
  - Research Site, Elizabethtown, Kentucky
  - Research Site, Crofton, Maryland
  - Research Site, Cumberland, Maryland
  - Research Site, Hagerstown, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Flowood, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Kalispell, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Manalapan, New Jersey
  - Research Site, Las Cruces, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Rochester, New York
  - Research Site, Roslyn, New York
  - Research Site, Syracuse, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Amarillo, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Mesquite, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Tacoma, Washington
- Canada (11):
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Bowmanville, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Reading
- Czechia (11):
  - Research Site, Brno
  - Research Site, Bruntál
  - Research Site, Česká Lípa
  - Research Site, České Budějovice
  - Research Site, Hlučín
  - Research Site, Liberec
  - Research Site, Ostrava - Trebovice
  - Research Site, Prague
  - Research Site, Sokolov
  - Research Site, Terezín
  - Research Site, Zlín
- Germany (3):
  - Research Site, Erlangen
  - Research Site, Hamburg
  - Research Site, München
- India (11):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Gandhinagar, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Lucknow
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Beer Yaakov
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Italy (4):
  - Research Site, Iesi, AN
  - Research Site, Legnano, MI
  - Research Site, Udine, UD
  - Research Site, Varese, VA
- Latvia (3):
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Valmiera
- Lithuania (3):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Šiauliai
- Portugal (3):
  - Research Site, Aveiro
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (4):
  - Research Site, Baia Mare
  - Research Site, Brailari
  - Research Site, Bucharest
  - Research Site, Ploieşti
- Serbia (4):
  - Research Site, Belgrade
  - Research Site, Kragujevac
  - Research Site, Niška Banja
  - Research Site, Novi Sad
- South Africa (6):
  - Research Site, Kempron Park, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Durban, Kz-natal
  - Research Site, Cape Town, W Cape
  - Research Site, Port Elizabeth
  - Research Site, Stellenbosch
- Spain (4):
  - Research Site, La Laguna (tenerife), Canary Islands
  - Research Site, Mérida, Extremadura
  - Research Site, Barcelona
  - Research Site, Getafe
- Ukraine (8):
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Simferopol
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhya
  - Research Site, Zaporyzhzhya
- United Kingdom (9):
  - Research Site, Maidstone, Kent
  - Research Site, Eastbourne, Sussex
  - Research Site, Solihull, West Midlands
  - Research Site, Basingstoke
  - Research Site, Cambridge
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Stoke-on-Trent
  - Research Site, Swindon

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=421&filename=CSR-D8480C00039.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1202&filename=CSR-D1700C00004.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=2264&filename=CSR-1939IL-0551.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1632 patients were enrolled: 308, 300 & 305 were randomised to Groups A, B & C, respectively (308, 298 & 302 received at least 1 dose of investigational product).
Pre-assignment Details: A total of 719 patients failed screening.
Groups:
- FOSTA 100 MG BID PO: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO: Dosing Group B
- PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO: Dosing Group C
Period: Overall Study
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Started | 308 (Patients who received treatment) | 298 (Patients who received treatment) | 302 (Patients who received treatment)
Randomised But Did Not Receive Treatment | 0 | 2 (Adverse event / Other) | 3 (Eligibility criteria not fulfilled / Severe non-compliance to protocol)
Completed | 174 (Number of patients who completed treatment includes patients who had a dose reduction.) | 168 (Number of patients who completed treatment includes patients who had a dose reduction.) | 129 (Number of patients who completed treatment includes patients who had a dose reduction.)
Not Completed | 134 | 130 | 173
Not completed — Not reported | 16 | 10 | 16
Not completed — Enrolment in long term extension | 57 | 66 | 119
Not completed — Severe non-compliance to protocol | 3 | 4 | 1
Not completed — Lack of therapeutic response | 9 | 4 | 9
Not completed — Dev. of study specific discont. criteria | 13 | 6 | 2
Not completed — Lost to Follow-up | 1 | 4 | 2
Not completed — Adverse Event | 35 | 36 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO | Total
Number analyzed (Participants) | 308 | 298 | 302 | 908
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.3) | 54 (11.6) | 53 (11.8) | 53 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 245 | 252 | 742
  Male | 63 | 53 | 50 | 166
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 254 | 235 | 241 | 730
  Black or African American | 6 | 15 | 8 | 29
  Asian | 16 | 13 | 20 | 49
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Indian or Pakistani | 25 | 31 | 28 | 84
  Other | 7 | 2 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With ACR20 at Week 24, Comparison Between Fostamatinib and Placebo
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, CRP = C-reactive protein, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: 24 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle.
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders | 39.6 | 39.6 | 24.5
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; Non-responder imputation has been applied following premature withdrawal, or increased dose of DMARD or any DMARD initiation, or for 8 weeks following receipt of any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — Week 24; Treatment difference in proportion of responders using a Mantel Haenszel approach stratified by background use of DMARD and pooled country; Weighted difference in proportions = 0.15, 95% CI 2-sided [0.08 to 0.22]

2. Secondary Outcome: Proportion of Patients Achieving ACR20, Comparison Between Fostamatinib and Placebo at Week 1
Description: as for outcome 1
Time Frame: 1 week
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Groups:
- FOSTA 100 MG BID PO (Combined): Dosing Group A and B combined
Arm/Group | FOSTA 100 MG BID PO (Combined) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 606 | 302
Percentage of responders | 16.0 | 8.3
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO (Combined) vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; 95% confidence intervals and p-values are calculated using a Mantel Haenszel approach stratified by background use of DMARD and pooled country; Weighted difference in proportion = 0.08, 95% CI 2-sided [0.04 to 0.12]

3. Secondary Outcome: Proportion of Patients Achieving ACR50, Comparison Between Fostamatinib and Placebo at Week 24
Description: ACR50: American College of Rheumatology 50% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, CRP = C-reactive protein, DMARD = Disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders | 20.8 | 18.1 | 8.3
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; [statistical method as in outcome 2, analysis 1]; Weighted difference in proportions = 0.13, 95% CI 2-sided [0.07 to 0.18]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; [statistical method as in outcome 2, analysis 1]; Weighted difference in proportions = 0.10, 95% CI 2-sided [0.05 to 0.15]

4. Secondary Outcome: Proportion of Patients Achieving ACR70, Comparison Between Fostamatinib and Placebo at Week 24
Description: ACR70: American College of Rheumatology 70% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as CRP) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, CRP = C-reactive protein, DMARD = Disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders | 9.1 | 6.0 | 2.6
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; [statistical method as in outcome 2, analysis 1]; Weighted difference in proportions = 0.07, 95% CI 2-sided [0.03 to 0.10]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.033, Mantel Haenszel; [statistical method as in outcome 2, analysis 1]; Weighted difference in proportions = 0.03, 95% CI 2-sided [0.00 to 0.07]

5. Secondary Outcome: ACRn - Comparison Between Fostamatinib and Placebo at Week 24
Description: ACRn: American College of Rheumatology index of RA improvement, based on smallest percentage improvement in the count of swollen joints (out of 28 joints), count of tender joints (out of 28 joints), or in blood test measures of inflammation (such as CRP) or the physician or patient's own assessments of disease activity, pain and physical function. Scores are reported as a percentage improvement on a scale of -100 to +100, with larger values representing a better clinical outcome. BID = twice daily, CI = confidence interval, CRP = C-reactive protein, DMARD = Disease-modifying anti-rheumatic drug, PO = orally, QD = once a day. Mean refers to change at Week 24.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage improvement from baseline
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage improvement from baseline | 20.75 (31.203) | 18.31 (28.427) | 9.84 (23.219)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Van Elteren — Nominal p-value presented for treatment comparison. Outcome was not formally tested within the predefined multiplicity procedure. As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; P-values are estimated using the Van Elteren test stratified by background use of DMARD and pooled country
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; Non-responder imputation has been applied following premature withdrawal, or increased dose of methotrexate or any DMARD initiation, or for 8 weeks following receipt of any parenteral steroids, or for patients with no post baseline data; Test type: Superiority or Other; p < 0.001, Van Elteren — [p-value comment as in outcome 5, analysis 1]; P-values are estimated using the Van Elteren test stratified by background use of DMARD and pooled country

6. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP <2.6 at Week 12, Comparison Between Fostamatinib and Placebo
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. A DAS28-CRP score of <2.6 is indicative of remission of RA symptoms. BID = twice daily, CRP = C-reactive protein, DMARD = Disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders | 17.2 | 10.7 | 3.0
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds ratio and 95% confidence intervals calculated using Logistic Regression with treatment, background use of DMARD and pooled country as factors; Odds Ratio (OR) = 7.1, 95% CI 2-sided [3.42 to 14.80] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 4.0, 95% CI 2-sided [1.88 to 8.65] — An odds ratio >1 indicates a benefit towards fostamatinib

7. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP <2.6 at Week 24, Comparison Between Fostamatinib and Placebo
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. A DAS28-CRP score of <2.6 is indicative of remission of RA symptoms. BID = twice daily, CRP = C-reactive protein, DMARD = Disease-modifying anti-rheumatic drug, OR=odds ratio, PO = orally, QD=once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders | 41.3 | 12.8 | 2.3
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 7.3, 95% CI 2-sided [3.23 to 16.65] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 6.4, 95% CI 2-sided [2.81 to 14.71] — An odds ratio >1 indicates a benefit towards fostamatinib

8. Secondary Outcome: Proportion of Patients Achieving DAS28 EULAR Response at Week 24
Description: Change in DAS28 was derived for each post baseline scheduled assessment and categorised using the European League Against Rheumatism (EULAR) response criteria. BID = twice daily, DAS28 = Disease Activity Score based on a 28-joint count, DMARD = disease-modifying anti-rheumatic drug, OR=odds ratio, PO = orally, QD = once a day.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders
  No response | 42.9 (1.46) [0.20 to 0.68] | 45.3 (1.34) [0.26 to 0.89] | 64.6 (1.30) [0.20 to 0.65]
  Moderate response | 33.8 | 34.9 | 29.1
  Good response | 23.4 | 19.8 | 6.3
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional odds model — Nominal p-value presented for treatment comparison. Outcome was not formally tested within the predefined multiplicity procedure; No Response, moderate response and good response are included in the model, with treatment, background use of DMARD and pooled country as factors; Odds Ratio (OR) = 2.84, 95% CI 2-sided [2.06 to 3.91] — An odds ratio > 1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional odds model — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 8, analysis 1]; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.77 to 3.37] — An odds ratio > 1 indicates a benefit towards fostamatinib

9. Secondary Outcome: HAQ-DI Response - Comparison of the Change(>=0.22) From Baseline Between Fostamatinib and Placebo at Week 24
Description: HAQ-DI: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is then calculated by summing the category scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygiene, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with a higher score indicating greater disability. The HAQ-DI response is a reduction from baseline in HAQ-DI score greater than or equal to the minimally important difference (0.22). BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Percentage of responders | 46.1 | 42.3 | 26.5
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.4, 95% CI 2-sided [1.73 to 3.46] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.46 to 2.94] — An odds ratio >1 indicates a benefit towards fostamatinib

10. Secondary Outcome: Change From Baseline to Week 24 in mTSS, Comparison Between Fostamatinib and Placebo
Description: mTSS: modified total sharp score, a measure of structural progression based upon X-rays. Hand and foot joints are scored for erosions and joint space narrowing and the results summed to give a value between 0 and 448. A higher value represents more serious progression of the disease. After disregarding ineligible records, patients with 2 or more non-missing values have had missing data imputed via linear extrapolation/interpolation methods. Patients with only 1 result were excluded from the analysis. ANCOVA = analysis of covariance, BID = twice daily, IP = investigational product, QD = once a day.
Time Frame: Baseline and 24 weeks
Population: The full analysis set includes patients who received at least 1 dose of IP. Patients were analysed by randomised treatment in accordance with the intention to treat principle. Measurements at 2 timepoints are required for a patient to be included in the analysis; therefore patients with only 1 result have been excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Units on a scale | 0.64 (3.130) | 0.37 (3.095) | 1.16 (5.849)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; This analysis is performed using an ANCOVA model on the ranks of the change from baseline, by pooled country and background use of DMARD, including a term for the ranks of the baseline score as a covariate; Test type: Superiority or Other; p = 0.904, Cochran-Mantel-Haenszel — As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; Residuals from ANCOVA are analysed using a Cochran-Mantel-Haenszel approach, adjusting for the effects of pooled country and background use of DMARD
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.342, Cochran-Mantel-Haenszel — As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: SF-36 - Comparison of the Change in PCS From Baseline Between Fostamatinib and Placebo at Week 24
Description: SF-36: 36-item Short Form Health Survey, a measure of health related quality of life. Scores for 8 sub-domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Function, Role-Emotional and Mental Health) are derived and normalised to a scale of 0-100. Physical and mental component scores (PCS and MCS) are derived by multiplying each of these 8 scores by a constant, summing them and standardising against a population with mean of 50+/- 10. Higher scores represent a better quality of life. Mean changes from baseline score are presented as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. ANCOVA = analysis of covariance, BID = twice daily, DMARD = disease modifying antirheumatic drugs, PO = orally, QD = once a day.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Units on a scale | 5 (7.2) | 4 (6.6) | 2 (5.7)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; Including terms for baseline as continuous covariate and treatment, background use of DMARD and pooled country as factors; Treatment difference = 2.47, 95% CI 2-sided [1.47 to 3.48]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 11, analysis 1]; Treatment difference = 1.64, 95% CI 2-sided [0.63 to 2.65]

12. Secondary Outcome: SF-36 - Comparison of the Change in MCS From Baseline Between Fostamatinib and Placebo at Week 24
Description: as for outcome 11
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO
Number analyzed (Participants) | 308 | 298 | 302
Units on a scale | 3 (7.5) | 3 (8.4) | 1 (6.3)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 11, analysis 1]; Treatment difference = 2.09, 95% CI 2-sided [0.97 to 3.20]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO (24 WKS) THEN FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 11, analysis 1]; Treatment difference = 1.96, 95% CI 2-sided [0.83 to 3.08]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: For placebo treated patients time frame includes both placebo (24 weeks) and fostamatinib (28 weeks) treatment. 11 SAEs occurred during the 24 week placebo treated period.
Groups:
- FOSTA 100 MG BID: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD: Dosing Group B
- PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period: Dosing Group C
Arm/Group | FOSTA 100 MG BID | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - Placebo Period
Serious Adverse Events (participants affected / at risk) | 30/308 | 25/298 | 10/302 | 10/302
Other Adverse Events (participants affected / at risk) | 170/308 | 152/298 | 42/302 | 77/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=308) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD (N=298) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=302) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=302)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MACULAR HOLE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HEPATOCELLULAR INJURY (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DENGUE FEVER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENTEROCOLITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS BACTERIAL (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
GASTROINTESTINAL BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OBESITY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
BONE NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
METASTATIC BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUMBAR RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UTERINE POLYP (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PULMONARY TOXICITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID (N=308) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD (N=298) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - FOSTA Period (N=302) | PLACEBO (24 WKS) THEN FOSTA 100 MG BID - Placebo Period (N=302)
DIARRHOEA (Gastrointestinal disorders) | 44 (44) | 47 (47) | 15 (15) | 13 (13)
NAUSEA (Gastrointestinal disorders) | 20 (20) | 17 (17) | 5 (5) | 7 (7)
NASOPHARYNGITIS (Infections and infestations) | 37 (37) | 29 (29) | 2 (2) | 16 (16)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 21 (21) | 14 (14) | 2 (2) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 17 (17) | 13 (13) | 3 (3) | 4 (4)
BLOOD PRESSURE INCREASED (Investigations) | 15 (15) | 15 (15) | 1 (1) | 10 (10)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 19 (19) | 23 (23) | 1 (1) | 10 (10)
HEADACHE (Nervous system disorders) | 19 (19) | 12 (12) | 5 (5) | 9 (9)
HYPERTENSION (Vascular disorders) | 68 (68) | 55 (55) | 17 (17) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less